CLINICAL TRIAL: NCT04850638
Title: Drug Interaction Between SHR4640 Tablets and Furosemide Tablets in Healthy Volunteers (Single Center, Single Arm, Open, Self-control)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR4640-108
Record Dates: First submitted 2021-04-19; First posted 2021-04-20 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — ruzinurad; Furosemide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR4640 tablets (Experimental)
  Interventions: Drug: SHR4640 tablets and furosemide tablets

INTERVENTIONS:
Drug: SHR4640 tablets and furosemide tablets — SHR4640 tablets and furosemide tablets

SUMMARY:
The purpose of this study was to evaluate the effect of SHR4640 tablets on the pharmacokinetics of furosemide tablets in healthy male volunteers, using a single-center, single-arm, open, self-control design.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the activities related to this trial, and be able to understand the procedures and methods of this trial, and be willing to strictly abide by the clinical trial plan to complete this trial;
2. Adult males aged between 18 and 45 (including both ends, whichever is the time of signing the informed consent form);
3. Body weight ≥ 50kg and body mass index (BMI): 19~26kg/m2 (including both ends).

Exclusion Criteria:

1. Have a fertility plan or refuse to use medically approved contraceptives within 1 month from the screening period to the last medication;
2. Smokers (those who smoke more than 5 cigarettes per day on average);
3. During the first month of screening, the average daily alcohol intake was more than 25g (for example, 750mL beer, 250mL wine, or 50mL liquor) or those who were positive for alcohol in blood test or alcohol breath test during screening;
4. Those who have eaten grapefruit or its fruit juice products, any caffeine (such as coffee, tea, chocolate, cola or other caffeinated carbonated drinks, etc.), alcoholic food or beverages within 2 days before administration;
5. Drug abusers or those who were positive in urine drug test during screening;
6. The researchers judged that the subjects had medical conditions that affected the absorption, distribution, metabolism and excretion of drugs or reduced compliance
7. Any clinical history of serious illness or any disease or condition that the researchers believe may affect the results of the trial, including, but not limited to, a history of circulatory, endocrine, nervous system, digestive, urinary or blood, immune, mental and metabolic diseases;
8. Allergic constitution, or allergic to any ingredient in SHR4640 and furosemide tablets, or allergic to sulfonamides or thiazide diuretics, or allergic to any food ingredient, or having special dietary requirements, unable to follow a uniform diet;
9. Previous history of urinary diseases (such as benign prostatic hyperplasia, urinary tract stenosis) or other diseases that lead to dysuria;
10. Screen those who have undergone any operation within the first 3 months, or who have not recovered after the operation, or who may have a plan for operation or hospitalization during the trial;
11. Those who donated blood (or lost blood) and donated blood (or lost blood) ≥ 400 mL within 3 months before screening, or received blood transfusion;
12. During screening, physical examination, vital signs, laboratory examination (whole blood cell analysis, blood biochemical analysis, blood electrolyte examination, urine analysis, fasting blood lipids, thyroid function), 12-lead ECG, X-chest X-ray and abdominal B-ultrasound were abnormal and had clinical significance.
13. When screening, systolic blood pressure was less than 90mmHg or greater than 140mmHg, and / or diastolic blood pressure was less than 60mmHg or greater than 90mmHg;
14. Urinary system ultrasound suggested or suspected urinary system crystals or stones during screening;
15. Those whose serum uric acid was higher than 420 μ mol / L or had a previous history of hyperuricemia and / or gout;
16. The level of serum potassium was lower than that of 4.0mmol/L during screening.
17. According to the serum creatinine within 2 weeks before administration, the glomerular filtration rate ((estimated glomerular filtration rate, eGFR) calculated by the simplified kidney disease diet adjustment (modification of diet in renal disease, MDRD) formula (Annex 1) is less than 90 mL/min/1.73 m ².
18. Those who were positive for hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody, or syphilis antibody within one month before the screening;
19. Screening people who have participated in any drug or medical device clinical trial within the previous 3 months (subject to signing informed consent);
20. Used any prescription drugs, over-the-counter drugs, Chinese herbal medicines or dietary supplements within 2 weeks before screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Cmax | Day1 to Day10
  Peak plasma concentration
AUC0-t | Day1 to Day10
  Area under the curve from the time of dosing. Dosing time to the last measurable (positive) concentration.
AUC0-inf (if available) | Day1 to Day10
  Area under the curve from time 0 to infinity
Ae | Day1 to Day10
  Cumulative Amount of excretion
CLr | Day1 to Day10
  Renal Clearance

SECONDARY OUTCOMES:
t1/2 | Day1 to Day10
  Half time
Tmax | Day1 to Day10
  Time of maximum observed concentration.
CL/F | Day1 to Day10
  apparent clearance
Vz/F | Day1 to Day10
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided